CLINICAL TRIAL: NCT03134768
Title: To Investigate the Immediate Effect of Birth on Immunological Parameters in Cord Blood, and Compare With Data of CS Born Infants Collected in the JULIUS SN Study
Brief Title: Effect of Birth on Immunological Parameters in Cord Blood
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAE.1C.D.10
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Immunologic Activity Alteration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — cord blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is not an interventional study — This is an observational study

SUMMARY:
The purpose of the study is to understand the immediate effect of birth on immunological parameters in vaginally born cord blood.

DETAILED DESCRIPTION:
The main purpose of the study is to understand the immediate effect of birth on immunological parameters in vaginally born cord blood and also whether mode and duration of delivery has an influence on immune parameters in cord blood.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers undergoing normal vaginal delivery

Exclusion Criteria:

* Use of non-steroidal anti-inflammatory drugs (NSAIDs) 2 weeks prior to birth

  * Antenatal antibiotics treatment (2 weeks prior to birth)
  * Diabetes mellitus requiring insulin treatment during pregnancy
  * Uncontrollable Hyperthyroidism during pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant mothers
Study Population: Pregnant mothers undergoing normal vaginal delivery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2017-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sandalova, PhD, Study Chair — Danone Asia Pacific Holdings Ltd; Anne Goh, MD, Study Chair — KK Hospital; Mei Chin Chua, MD, Principal Investigator — KK Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in KK Women's and Children's Hospital
Groups:
- Vaginally Born Children: Cord blood samples collected from vaginally born children
Period: Overall Study
Arm/Group | Vaginally Born Children
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vaginally Born Children
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 0 [0 to 0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Cytokines Profile in Cord Blood Plasma
Description: Following cytokines will be part of the profile: IL-6, IL-1, IL-2, IL-4, IL-5, IL-7, IL-8, IL-10, IL12p70, IL-13, IL-17, G-CSF, GM-CSF, IFNg, MCP-1(MCAF), MIP-1b, TNFa
Time Frame: 1 year
Population: Other cytokines were out of detection limits.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vaginally Born Children
Number analyzed (Participants) | 50
pg/ml
  IL-6 | 1.6 (7.1)
  TNFa | 21.81 (8.4)
  IL-8 | 165 (279)
  G-SCF | 14 (44)

2. Primary Outcome: Cord Blood Immunoglobulin Levels
Description: Immunoglobulin levels will be measured in cord blood plasma
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vaginally Born Children
Number analyzed (Participants) | 50
pg/ml
  IgE | 1.7 (2)
  IgG | 2613064 (3066008)

3. Primary Outcome: Allergen Stimulated Cytokine Expression in the Supernatants of Cord Blood Mononuclear Cells (CBMC)
Description: Cellular response to allergen stimulation will be measured in supernatants of cultured cord blood mononuclear cells.
Time Frame: 1 year
Population: IL-6 was measured after incubation with House Dust mite extracts. The mean expression of IL-6 by the cord blood mononuclear cells in response to house dust mite extract is presented here.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vaginally Born Children
Number analyzed (Participants) | 50
pg/ml | 18612 (38892)

ADVERSE EVENTS:
Arm/Group | Vaginally Born Children
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less